CLINICAL TRIAL: NCT03651414
Title: Safety Issues and SurvIval For Medical Outliers (SISIFO) - Not-for-profit Observational Study to Evaluate the Quality and Safety of Care in Patients "Outliers" Hospitalized With Medical Diseases
Brief Title: Safety Issues and SurvIval For Medical Outliers
Acronym: SISIFO
Status: Terminated | Type: Observational
Why Stopped: Due to health emergency Covid-19.
Sponsor: Fadoi Foundation, Italy (Other)
Collaborators: University of Genova (Other)
Responsible Party: Sponsor
Other Study IDs: FADOI.08.2018
Record Dates: First submitted 2018-08-24; First posted 2018-08-29 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Hospitalization
Keywords: Outliers

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: Patients hospitalized ab initio in Internal Medicine or similar for at least one night
  Interventions: Other: Clinical data collection
- Outlier: Patients spending at least one night in a ward different from Internal Medicine despite the presence of medical diseases, due to lack of available beds
  Interventions: Other: Clinical data collection

INTERVENTIONS:
Other: Clinical data collection — There will not be any experimental intervention. The study will be conducted according with normal clinical practice.

SUMMARY:
Each Investigator will have to record data concerning 70 patients. In particular 40 patients "outliers" and 30 patients "control".

DETAILED DESCRIPTION:
Phase 1 - Patients enrollment (October 2018 - May 2019) Each Investigator will have to record data concerning 70 patients. In particular 40 patients "outliers" (max 10 per month) and 30 patients "control" (max 6 per month). It will be collected clinical and organisational information. The Investigators of the wards that will not have patients "outliers" will have to enroll 70 patients "control" (max 15 per month).

Phase 2 - Database review and validation (June 2019 - October 2019) The data collected will be analysed to process the endpoints.

ELIGIBILITY:
Inclusion Criteria:

Outlier:

* Age ≥ 18 years
* Signature of informed consent
* Patients coming from Emergency Room
* Patients to be hospitalized in Internal Medicine or similar (not day-hospital)
* Patients spending at least one night in another ward for lack of available beds
* Consecutive cases

Control:

* Age ≥ 18 years
* Signature of informed consent
* Patients coming from Emergency Room
* Patients to be hospitalized in Internal Medicine or similar (not day-hospital)
* Patients hospitalized ab initio in Internal Medicine or similar for at least one night
* Consecutive cases

Exclusion Criteria (Outlier and Control):

* Age < 18 years
* Patients hospitalized in Internal Medicine or similar coming from other wards or directly from home

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized for any cause.
Sampling Method: Non-Probability Sample
Enrollment: 2056 (Actual)
Dates: Start 2018-10-19 (Actual); Primary Completion 2020-04-07 (Actual); Study Completion 2020-07-07 (Actual)

PRIMARY OUTCOMES:
Inhospital mortality | 8 months
  Evaluation of the inhospital mortality in patients "outliers" compared to patients that are hospitalized ab initio in the relevant ward (Internal Medicine - patients "control")

SECONDARY OUTCOMES:
Adverse Events | 8 months
  Evaluation of the adverse events in patients "outliers" compared to patients that are hospitalized ab initio in the relevant ward (Internal Medicine - patients "control")
Mortality rate | 3 months
  Mortality rate after 30 days and after 3 months from the hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Mauro Campanini, Study Director — FADOI Foundation
Locations (32):
- Italy (32):
  - Ospedale di Bisceglie - Trani, Bisceglie
  - Azienda Ospedaliera Brotzu, Cagliari
  - Ospedale Santissima Trinità, Cagliari
  - Ospedale Cervesi, Cattolica
  - Ospedale di Conegliano, Conegliano
  - Istituti Ospitalieri di Cremona, Cremona
  - Ospedale Morgagni Pierantoni, Forlì
  - Ospedale Evangelico, Genova
  - Ospedale Policlinico S. Martino, Genova
  - Ospedale Villa Scassi, Genova
  - Ospedale Sant'Andrea, La Spezia
  - Ospedale S. Maria Goretti, Latina
  - Ospedale di Lavagna, Lavagna
  - Ospedale di Legnano, Legnano
  - Ospedale di Magenta, Magenta
  - Ospedale San Carlo Borromeo, Milan
  - Ospedale Buon Consiglio Fatebenefratelli, Napoli
  - Ospedale Felice Lotti, Pontedera
  - Nuovo Ospedale S. Stefano, Prato
  - Ospedale Infermi, Rimini
  - Ospedale San Giovanni Calibita Fatebenefratelli, Roma
  - Ospedale San'Antonio, San Daniele del Friuli
  - Ospedale Nostra Signora di Bonaria, San Gavino Monreale
  - Ospedale G. Borea, Sanremo
  - Ospedale San Bartolomeo, Sarzana
  - Ospedale Civile SS Annunziata, Sassari
  - Ospedale di Sestri Levante, Sestri Levante
  - Azienda Ospedaliera S. Maria, Terni
  - Ospedale Cottolengo, Torino
  - Ospedale di Treviglio, Treviglio
  - Ospedale Sant'Andrea, Vercelli
  - Ospedale Civile di Voghera, Voghera